CLINICAL TRIAL: NCT03277898
Title: Aerobic Exercise and Cognitive Functioning in Women With Breast Cancer: the ACTIVATE Trial
Brief Title: Aerobic Exercise and Cognitive Functioning in Women With Breast Cancer
Acronym: ACTIVATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Cancer Society (CCS) (Other); Avon Foundation (Other); University of Ottawa (Other); British Columbia Cancer Agency (Other)
Responsible Party: Principal Investigator, Kristin Campbell, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H17-00563
Record Dates: First submitted 2017-08-03; First posted 2017-09-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Breast Neoplasms
Keywords: Breast Neoplasms; Exercise* OR "Aerobic Exercise"; Cognitive Function*; "Antineoplastic therapy" OR "Antineoplastic agent"; Chemotherapy, Adjuvant; Chemotherapy, Neoadjuvant
MeSH Terms: conditions — Breast Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise (Experimental): Participants will complete three supervised aerobic exercise sessions each week using the treadmill, stationary bicycle or elliptical training for the duration of their chemotherapy (12-18 weeks). Aerobic exercise will be performed for 20-40 minutes at 50-75% of heart rate reserve. Participants will wear heart rate monitors during all supervised sessions (Polar Electro Inc., Lake Success, NY) and will be provided with target heart rates that will be individualized using their baseline (i.e., week 0) assessment data. Home-based exercise will be introduced in week 3. For the home-based sessions, participants will be asked to complete at least 1 session per week of 30 minutes of aerobic exercise (an activity of their choosing; e.g., walking).
  Interventions: Behavioral: Aerobic Exercise
- Usual Care (Wait-list Control) (Other): Participants randomly assigned to UC group will be advised to continue with their regular activities of daily living. Following their chemotherapy, the UC group will receive the exercise intervention (lasting 12 weeks).
  Interventions: Behavioral: Usual Care (Wait-list Control)

INTERVENTIONS:
Behavioral: Aerobic Exercise — Three weekly moderate-vigorous intensity supervised aerobic exercise training for the duration of adjuvant chemotherapy. Home-based exercise will also be introduced in week 3 of the intervention.
  Arms: Aerobic Exercise
Behavioral: Usual Care (Wait-list Control) — Three weekly moderate-vigorous intensity supervised aerobic exercise training starting upon adjuvant chemotherapy completion. Home-based exercise will also be introduced in week 3 of the intervention.
  Arms: Usual Care (Wait-list Control)

SUMMARY:
In Canada, approximately 68 women are diagnosed with breast cancer every day. Chemotherapy-related cognitive changes (CRCC) are reported by up to 75% of breast cancer survivors during treatment and symptoms persist in 35% of survivors after treatment. Women report that CRCC negatively impacts their everyday functioning and substantially reduces their overall quality of life. Effective clinical interventions to manage CRCC are elusive. As a result, breast cancer survivors typically receive little to no advice on how to prevent or manage CRCC. Aerobic exercise is a type of physical activity that uses large muscle groups, is rhythmic in nature, and can be sustained for at least 10 minutes (e.g., walking, jogging, indoor cycling). It has been associated with improved quality of life in breast cancer survivors. It also holds great promise as an intervention to prevent or mitigate CRCC. However, there is limited evidence from experimental studies to confirm this. Therefore, the primary aim of this trial is to evaluate the impact of a supervised aerobic exercise intervention on CRCC in women diagnosed with early-stage breast cancer. Recruited women will be randomized into one of two groups: (1) aerobic exercise during chemotherapy, or (2) usual care during chemotherapy and the aerobic exercise post-chemotherapy (i.e., wait-list control group). This study will test several novel hypotheses, including whether exercise during chemotherapy can prevent and/or mitigate CRCC and its negative impact on quality of life among women with breast cancer, and whether the timing of the exercise intervention matters (i.e., exercise during versus after chemotherapy). The results of this study aim to address the concerns of women affected by CRCC who are currently lacking available evidence-based treatment options, as well as oncology care providers' need to have options to recommend to their patients to prevent or manage CRCC.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the impact of an aerobic exercise intervention on CRCC in women diagnosed with breast cancer who undergo chemotherapy. The specific objectives are to:

1. Test the effect of aerobic exercise during chemotherapy (EX) compared to a usual care wait-list control group (exercise after chemotherapy; UC) on CRCC as assessed by neuropsychological tests and self-report;
2. Test the effect of EX compared to UC on:

   1. Global measures of brain structure and functioning including brain volume in regions associated with working memory and response inhibition, white matter integrity (i.e., fractional anisotropy, mean diffusivity), and neural functioning using magnetic resonance imaging (MRI);
   2. Overall global brain network organization and improved regional brain network organization and neural functioning in areas underlying attention and working memory (i.e., dorso-lateral prefrontal cortex, superior temporal region and posterior parietal cortex) using electroencephalography (EEG; Vancouver site only; see Methods).
3. Assess if the timing of the exercise intervention (i.e., during chemotherapy versus after chemotherapy) moderates the effects on CRCC by examining the effects of the intervention at 1-year post start of chemotherapy.

It is hypothesized that:

1. At the end of chemotherapy, EX group will perform better than UC group on neuropsychological tests and will self-report better cognitive functioning;
2. At the end of chemotherapy, EX group will have maintained measures of brain structure and functioning as assessed by MRI scans and EEG (Vancouver site only) compared to UC group who will have significant changes in both;
3. At 1-year post the start of chemotherapy, EX group will have better outcomes compared to the UC group.

This is a two-arm, two-centre RCT. The two arms are:

1. Aerobic exercise intervention during chemotherapy (EX);
2. Usual care during chemotherapy and aerobic exercise after chemotherapy (i.e., usual care wait-list control group; UC).

Recruitment:

84 women diagnosed with breast cancer will be recruited across the two sites. The primary method of recruitment will be through printed postings and oncologist referral at the two main clinical sites: British Columbia Cancer Agency-Vancouver (BCCA) and The Ottawa Hospital (TOH). We anticipate our target of 84 patients will be reached in 30 months (combined site rate of 2-3 participants per month).

Outcomes will be assessed at:

1. Pre-chemotherapy (baseline, week 0);
2. Mid-chemotherapy (approximately 6-9 weeks post-baseline);
3. End of chemotherapy (approximately 12-18 weeks post-baseline);
4. Follow-up and post-usual care wait-list control group receiving the intervention (approximately 24-34 weeks post-baseline);
5. 1-year follow-up (52 weeks post-baseline).

Optional neuroimaging and EEG will be completed in a sub-set of participants at each site who are interested, eligible, and consent to additional assessments at these time points:

1. Pre-chemotherapy (baseline, week 0);
2. End of chemotherapy (approximately 12-18 weeks post-baseline);
3. 1-year follow-up (52 weeks post-baseline).

Intervention:

After obtaining informed consent, each participant will be scheduled for a baseline assessment (week 0). After baseline assessments, participants will be randomized. For the EX group, the intervention will be delivered concurrent with participants' chemotherapy regimen (lasting approximately 12-18 weeks). The intervention will be progressive aerobic exercise. The intervention is based on prior protocols used by the study team among women during treatment or who have completed treatment. Participants will complete three supervised 20-40 minute aerobic exercise sessions each week. Home-based exercise will be introduced in week 3. For the home-based sessions, participants will be asked to complete at least 1 session per week of 30 minutes of aerobic exercise (an activity of their choosing; e.g., walking).

Data Analysis:

Changes in objective and self-reported cognitive functioning will be analyzed based on repeated measures analysis of variance with fixed terms for treatment, time, and a treatment by time interaction. Clinically important baseline differences between the study arms will be included as covariates in all analyses. Correlation in repeated measures on the same individual over time will be accounted for by explicitly modeling the covariance matrix, with the best-fitting covariance structure decided using likelihood ratio tests and information criteria. The difference between the experimental and control arms at end of chemotherapy (primary comparison) will be calculated as adjusted least square mean difference in change from baseline, together with 95% confidence intervals. All tests will be evaluated at the two-sided 5% level of significance. SAS v.9.3 will be used for all analyses. Additional adjusted analyses will be carried out using potential covariates.

To explore changes in brain structure and functioning, data will be analyzed with SPM12 (VBM and CONN toolboxes) and FSL (FMRIB Software Library v5.0). Following respective post-processing procedures, pre- and post- intervention measurement comparisons will be conducted using voxel-wise statistical repeated-measures analyses, appropriate to each MRI technique (for example, FA, MD for the DTI data, seed-to-voxel functional connectivity for the fMRI data, as well as both whole brain and region of interest analyses of each fMRI task). Statistical maps will be inspected at p < 0.05 levels, corrected for multiple comparisons. To test the effect of aerobic exercise during chemotherapy compared to post-chemotherapy on outcomes 1-year after enrolment, the models as described above will additionally include the response at 1-year follow-up and the contrast of interest will be the difference in change from baseline (week 0) to 1-year post start of chemotherapy (week 52).

The sustainability of the intervention will be examined in each arm by testing the change in response from immediately post-intervention to week 52, together with a 95% confidence interval.

EEG signal processing will be completed using EEG time series from 27 locations to construct the brain connectivity networks. The network graphs will be computed for each subject using the false discovery rate controlled PC (PCFDR) algorithm, which is a statistical model that tests the conditional dependence/independence between any two regions based on all other brain regions. Partial correlation will be used to evaluate the conditional independence, which estimates the directed interactions between any two brain regions after removing the effects of all other brain areas. The FDR threshold will be set at a 5% level. Graph Theory Analysis will use the "Brain Connectivity Toolbox" running Matlab (Natick, MA) to carry out the graph theoretical based analysis. Traditional graph theoretical calculations will be used to characterize different features of the network of interest such as density, global efficiency, modularity and small-worldness.

Justification:

CRCC, or "chemo brain", is common among women diagnosed with breast cancer, significantly impacts everyday life, and diminishes quality of life. Women with breast cancer described their chemo brain symptoms as "frustrating", "upsetting" and for some "frightening". In addition, women with breast cancer may be unable to return to their previous occupational, family and social activities, or do so only with significant additional mental effort. As a result the high prevalence of chemo brain in women with breast cancer has a large economic burden due to demand of health care resources and lost work-force productivity. Women with breast cancer also report a general frustration in the response of the medical community, either due to lack of acknowledgement of their symptoms or the fact that intervention strategies are limited. Furthermore, there is limited information to guide health care professionals with regards to clinical guidelines for the management of chemo brain and health care professionals report that they do not consider themselves adequately knowledgeable to address chemo brain.

This study will test if exercise during chemotherapy can mitigate chemo brain and its negative impact on quality of life among women diagnosed with breast cancer, which if shown to be effective, will have profound effects on the lives of those with chemo brain as well as their family members and clinicians who currently have a lack of treatment options available.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with stage I-III breast cancer;
* Scheduled to receive adjuvant or neoadjuvant chemotherapy;
* Able to speak and understand English in order to complete the study outcome measures;
* Approval of medical oncologist to participate in the exercise intervention

Exclusion Criteria:

* Having previously received chemotherapy or radiation therapy;
* Score <24 at baseline on the Montreal Cognitive Assessment (MoCA; indicating moderate to severe cognitive impairment);
* Having received a diagnosis of severe anxiety or mood disorder within the past year;
* Having a medical condition that could impact cognition (e.g., prior head injury, substance use disorder);
* Currently meeting American College of Sports Medicine (ACSM) aerobic exercise guidelines for cancer survivors in the 3 months prior to enrolment;
* Body mass index ≥45 kg/m2;
* Mobility issues that require a mobility aid or that prevent exercise on a bike, treadmill, or elliptical (e.g., orthopedic injury, severe arthritis).

Additional Inclusion/Exclusion Criteria: During the screening process, patients will be informed that they can participate in additional optional assessments (i.e., MRI and EEG (Vancouver site only for EEG)

Additional inclusion criteria for MRI:

* Right-handedness, because language is lateralized and has been shown to be left side dominant (for right handers) during MRI tasks;
* Able to read, understand, and provide informed consent in English for the additional assessments.

Additional exclusion criteria for MRI are:

* Metal implants (e.g., pacemaker) or metal dental work (aside from fillings) that would preclude scanning;
* Claustrophobia;
* Poor eyesight (not correctable with contact lenses) that precludes viewing stimuli presented in the scanner;
* Lower back pain that would preclude a person from lying relatively still for one hour;
* Breast tissue expander(s) inserted in the surgery site.

Ages: 19 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Change with treatment and maintenance post-treatment in objective neuropsychology test battery composite score | Pre-chemotherapy (baseline, week 0), end of chemotherapy (12-18 weeks post-baseline), follow-up/post-usual care group receiving intervention (24-34 weeks post-baseline), 1-year follow-up (52 weeks post-baseline)
  A neuropsychological test battery. The tests are as follows: WAIS-IV (Digit-Symbol Coding, Letter-Number-Sequencing), Auditory Consonant Trigrams Test, Brief Visuospatial Memory Test Revised, Controlled Oral Word Association Test, Hopkins Verbal Learning Test-Revised, and Trail Making Test A&B. Alternate forms will be used, with the exception of the WAIS-IV tests, the Controlled Oral Word Association Test, and Trail Making A&B. These tests are combined to form a composite score called the COGSUM.

SECONDARY OUTCOMES:
Change with treatment and maintenance post-treatment in self-reported cognitive function and impact on quality of life | Pre-chemotherapy (baseline, week 0), mid-chemotherapy (week 6-9), end of chemotherapy (12-18 weeks post-baseline), follow-up/post-usual care group receiving intervention (24-34 weeks post-baseline), 1-year follow-up (52 weeks post-baseline).
  The Functional Assessment of Cancer Therapy (FACT)-Cognitive (Cog) Version 3
Change with treatment and maintenance post-treatment in self-reported cognitive function | Pre-chemotherapy (baseline, week 0), mid-chemotherapy (week 6-9), end of chemotherapy (12-18 weeks post-baseline), follow-up/post-usual care group receiving intervention (24-34 weeks post-baseline),1-year follow-up (52 weeks post-baseline).
  The Patient-Reported Outcomes Measurement Information System Applied Cognition short form
Change with treatment and maintenance post-treatment in brain function and structure | Pre-chemotherapy (baseline, week 0), end of chemotherapy (12-18 weeks post-baseline), 1-year follow-up (52 weeks post-baseline).
  Magnetic resonance imaging (MRI) assessment including a resting state fMRI procedure, a diffusion tensor imaging sequence, and three fMRI tasks (i.e., Letter N-Back and Word List Recognition Task).
Change with treatment and maintenance post-treatment in electrical activity of the brain | Pre-chemotherapy (baseline, week 0), end of chemotherapy (12-18 weeks post-baseline), 1-year follow-up (52 weeks post-baseline).
  Electroencephalogram (EEG) will be performed including five minutes of resting data and 20 minutes during a computerized task.

OTHER OUTCOMES:
Change with treatment and maintenance post-treatment in aerobic fitness | Pre-chemotherapy (baseline, week 0), end of chemotherapy (12-18 weeks post-baseline), follow-up (24-34 weeks post-baseline; UC participants only), 1-year follow-up (52 weeks post-baseline).
  Aerobic capacity (VO2peak) will be measured with a maximal cardiopulmonary test using a metabolic cart (PARVO Medics).
Change with treatment and maintenance post-treatment in resting blood pressure | Pre-chemotherapy (baseline, week 0), end of chemotherapy (12-18 weeks post-baseline), follow-up (24-34 weeks post-baseline; UC participants only), 1-year follow-up (52 weeks post-baseline).
  Resting blood pressure (mmHg), measured in duplicate on non-surgical side using a blood pressure monitor.
Change with treatment and maintenance post-treatment in body composition | Pre-chemotherapy (baseline, week 0), end of chemotherapy (12-18 weeks post-baseline), follow-up (24-34 weeks post-baseline; UC participants only), 1-year follow-up (52 weeks post-baseline).
  Height (using a stadiometer) and weight (using a standard scale)
Socio-demographic information | Pre-chemotherapy (baseline, week 0)
  Brief self-reported socio-demographic
Medical characteristics | Through study completion, an average of 1 year
  Measures will be extracted from participants' medical records at the Vancouver-BCCA and TOH (as appropriate). In particular, the following medical information will be extracted: cancer disease stage, treatment factors (i.e., type, timing, and dosage of all treatments including surgery/ies and adjuvant treatment(s)), and list of prescribed medications
Change in exercise behaviour | Pre-chemotherapy (baseline, week 0), end of chemotherapy (12-18 weeks post-baseline), follow-up and post-usual care wait-list control group receiving the intervention (24-34 weeks post-baseline), and 1-year follow-up (52 weeks)
  Modified version of the Leisure Time Exercise Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kristin L Campbell, PhD, Principal Investigator — Department of Physical Therapy
Locations (3):
- Canada (3):
  - Breast Cancer Training Center, 614 W. 8th Ave, Vancouver, British Columbia
  - Clinical Exercise Physiology Lab, Vancouver, British Columbia
  - School of Human Kinetics - University of Ottawa, Ottawa, Ontario

REFERENCES:
- [Derived] Damji S, Sattari S, Zadravec K, Campbell KL, Brunet J, Virji-Babul N. Changes in EEG Microstate Dynamics and Cognition Post-Chemotherapy in People With Breast Cancer. Brain Behav. 2025 Mar;15(3):e70335. doi: 10.1002/brb3.70335. PMID 40038798
- [Derived] Brunet J, Barrett-Bernstein M, Zadravec K, Taljaard M, LeVasseur N, Srikanthan A, Bland KA, Collins B, Kam JWY, Handy TC, Hayden S, Simmons C, Smith AM, Virji-Babul N, Campbell KL. Study protocol of the Aerobic exercise and CogniTIVe functioning in women with breAsT cancEr (ACTIVATE) trial: a two-arm, two-centre randomized controlled trial. BMC Cancer. 2020 Jul 31;20(1):711. doi: 10.1186/s12885-020-07196-3. PMID 32736542